CLINICAL TRIAL: NCT01489137
Title: The EC90 of Remifentanil Blunting Hemodynamic Changes to Head Fixation in the Patients Undergoing Neurosurgery
Brief Title: The EC90 of Remifentanil Blunting Hemodynamic Changes to Head Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_fixation_remifentanil
Record Dates: First submitted 2011-12-05; First posted 2011-12-09 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Brain Tumor; AVM; ICH
MeSH Terms: conditions — Brain Neoplasms | interventions — Remifentanil

ARMS (1):
- neurosurgery with fixation (Experimental)
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil — According to previous patient's response, the investigators will allocate the effect site concentration of remifentanil of next patient during head fixation. And, For this allocation of dose of remifentanil the investigators use biased coin design up-and-down method.
  For the first patient, the dose of remifentanil would be fixed at 5.5ng/ml which we predict as EC90. And, step size of dose is 0.5ng/ml.
  Other Names: Biased coin design up-and-down method.

SUMMARY:
The purpose of this study is to estimate the EC90 of remifentanil blunting hemodynamic changes to head fixation in the patients undergoing neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing neurosurgery that require head fixation with mayfield head holder
* patients who agree to our study

Exclusion Criteria:

* patients who don't agree to our study
* BMI<16.0 or BMI>30
* cardiovascular disease, pulmonary disease, renal disease
* alcoholic abuser or drug abuser
* patients who takes any drug having an influence on cardiovascular system or sympathetic nervous system
* any use of local anesthetics or drugs which have an influence on cardiovascular system from beginning of induction to peri-fixation period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
mean arterial blood pressure | peri-fixation periord
  mean arterial blood pressure will be recorded at 2 minutes before fixation, 1 minute before fixation, highest value during immediately post-fixation periord, 1 minute after fixation, 2 minutes after fixation, 3 minutes after fixation, 4 minutes after fixation and 5 minutes after fixation.
heart rate | peri-fixation periord
  heart rate will be recorded at 2 minutes before fixation, 1 minute before fixation, highest value during immediately post-fixation periord, 1 minute after fixation, 2 minutes after fixation, 3 minutes after fixation, 4 minutes after fixation and 5 minutes after fixation.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee JM, Bahk JH, Lim YJ, Lee J, Lim L. The EC90 of remifentanil for blunting cardiovascular responses to head fixation for neurosurgery under total intravenous anesthesia with propofol and remifentanil based on bispectral index monitoring: estimation with the biased coin up-and-down sequential method. BMC Anesthesiol. 2017 Oct 10;17(1):136. doi: 10.1186/s12871-017-0426-z. PMID 29017455